CLINICAL TRIAL: NCT01073683
Title: Phase II Organ Preservation Trial Using Cisplatin Concomitant With Radiation Therapy in Advanced Laryngeal Cancer Patients Who Have Responded to Induction Chemotherapy With Taxotere, Cisplatin, and 5-Fluorouracil (TPF)
Brief Title: Induction Docetaxel/Cisplatin/5-fluorouracil (TPF) as Selector for Chemo Radiation Therapy (RT) Versus Partial Laryngectomy in Advanced Laryngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Davidoff Cancer Center (Unknown)
Responsible Party: Aron Popovtzer senior doctor, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC5476
Record Dates: First submitted 2010-01-12; First posted 2010-02-23 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-02

CONDITIONS: Larynx Cancer
Keywords: TPF; INDUCTION CHEMOTHERAPY; LARYNX PRESERVATION; SUPACRICOID LARYNGECTOMY; Stage 3 and 4 larynx cancer
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Laryngoscopy; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- larynx preservation (Experimental): Decision between surgery and Chemo-rt according to response to initial induction chemotherapy
  Interventions: Procedure: laryngoscopy; Drug: Taxotere (Docetaxel), Cisplatin, 5FU

INTERVENTIONS:
Procedure: laryngoscopy — Treatment of advanced larynx cancer with induction TPF, in order to decide between chemoradiation and laryngeal preservation surgery
  Other Names: supracrocoid laryngectomy
Drug: Taxotere (Docetaxel), Cisplatin, 5FU — Taxotere 75 mg/m2 D1, Cisplatin 75 mg/m2 D1, 5FU 750 mg/m2 D1-4

SUMMARY:
Treatment of patients with one cycle of induction chemotherapy to select for organ preservation of the larynx has been proven as a standard approach. When compared to historical controls. The investigators propose to study patients with a similar treatment strategy (i.e. one cycle of induction chemotherapy followed by two more chemotherapy cycles, in advanced nodal disease, followed by chemoradiation for those responding to the initial chemotherapy. Those who fail to respond or fail in radiation will directly undergo surgery. The novelty of the proposed study is that non responders and failures will be given the opportunity of larynx preserving supracricoid laryngectomy. The investigators will attempt to reduce toxicity from induction chemotherapy and improve potency with the use of docetaxel/cisplatin/5-fluorouracil (TPF) in place of the standard regimen of cisplatin and 5-fluorouracil (PF). Emerging data demonstrates that induction regimens containing triplets with platinum, 5-fluorouracil, and taxanes produce higher response rates and less overall toxicity when compared to induction strategies utilizing PF

DETAILED DESCRIPTION:
The optimal treatment of patients with laryngeal cancer remains controversial. Standard treatment options have included laryngectomy with or without radiation (RT) and radiation alone with surgical salvage (RTSS).

Because of the significant functional morbidity associated with laryngectomy, the Department of Veterans Affair Cooperative Studies Program completed a randomized, prospective study of 332 patients that compared a new organ preservation treatment strategy to conventional laryngectomy and radiation. The experimental treatment arm involved three cycles of neoadjuvant chemotherapy followed by definitive radiation among patients who had a partial (>50%) clinical tumor response. Final results of this study demonstrated comparable 2, 3, 4, and 10 year survival rates between treatment groups, with successful laryngeal preservation in 66% of the surviving patients randomized to receive neoadjuvant chemotherapy.

This study led to a dramatic re-assessment of the treatment approach for advanced laryngeal and hypopharyngeal cancer patients, who face total laryngectomy. Based on these results, Second approach was designed and tested in a Phase II study at the University of Michigan .In this study, 97 patients were treated with one cycle of induction chemotherapy. Seventy-five percent had a >50% reduction of tumor and were treated with chemo-RT (cisplatin 100 mg/m2 x 3 cycles), and 25% were non-responders who underwent total laryngectomy followed by RT. The overall 3-year survival rate was 85%,and the larynx preservation rate was 70%. This study included over 30 percentage of patients with advanced stage 4 disease, however did not specifically evaluate there outcome and therefore did not directly address the role of organ preservation in advanced disease which is considered a controversial issue in head and neck literature.

In this study all patients (25 %) who did not respond to the initial chemotherapy were referred to total laryngectomy and therefore there were 30 %of patients who eventually underwent total laryngectomy.Lately several series suggest the option of partial laryngectomy as an alternative to total laryngectomy as initial treatment for advanced larynx cancer ,in cases in which the cricoids cartilage and arytenoids are not involved.Supracricoid subtotal laryngectomy spares at least one arytenoid and offers organ preservation and can also be performed according to many articles as salvage surgery in cases of radiation failure,and therefore if performed in the right indications can improve the percentage of total laryngectomy free patients without compromising survival. This will reflect of course on quality of life It has been suggested lately that the use of aggressive induction chemotherapy may improve outcome. The combination of Taxotere with Cisplatin and 5-fluorouracil has been shown to be more effective than the standard cisplatin and 5-fluorouracil without an elevation in side effects .It has been suggested that the three cycles of induction chemotherapy may lower the rate of distant metastases which is high in advanced disease

Objectives

Primary

To determine the laryngeal preservation rate in a treatment paradigm that uses clinical response to a single cycle of induction chemotherapy to select patients for either concurrent cisplatin-radiation or surgery(if possible organ preserving partial laryngectomy) as compared to historical controls To determine the survival rate among T4 laryngeal patients in a treatment paradigm that uses clinical response to a single cycle of induction chemotherapy to select patients to either ,two more cycles of induction followed by concurrent cisplatin-radiation or surgery .

Secondary To determine the survival rate in a treatment paradigm that uses clinical response to a single cycle of induction chemotherapy to select patients for either concurrent cisplatin-radiation or surgery including organ preserving partial laryngectomy (if possible) as compared to historical controls.

To determine if the use of three cycles of induction chemotherapy lowers the rate of distant metastases in advanced cases; namely: positive nodal disease and T4.

To evaluate the quality of life (QOL) of this treatment paradigm.

To evaluate partial supracricoid laryngectomy as salvage to chemoradiation failure.

compare PET scan results with the pathological specimen of the larynx.

To determine correlation between changes in biological markers such as EGFR degradation EGFR mutation, p53 overexpression, Bcl-XL, Bcl-2 expression, and HPV observed in tumor biopsies taken shortly after the administration of TPF, compared with pre-treatment biopsies. And compared to those found in the completion of treatment in cases of failures.

Study Design

Chemotherapy/Radiation/Surgery schedule Days #1-4: Patients will undergo induction chemotherapy with (TPF) docetaxel (Taxotere) 75 mg/m2 and cisplatin 100 mg/m2 on day 1, and 5-FU CI 750mg /m2 /24 hours days 1-4. See section 7.2.

Day #22: Patients will undergo a direct laryngoscopy with biopsy the biopsy will be done with in 3 days. Patients will also undergo a repeat CT scan of the neck within a week (+/-) of their perspective biopsies.

Patient with a < 50% response (NR) to induction chemotherapy will undergo salvage supracricoid partial laryngectomy if possible or laryngectomy followed by RT. Cisplatin will be added to radiation for patients whose surgical pathology reveals high-risk features (i.e. extracapsular spread, > 2 positive lymph nodes, perineural invasion, or positive margins). Cisplatin will be dosed 35 mg/m2 weekly at the discretion of the prescribing physician. See section 7.2 for prescribing details for cisplatin.

Responding patients with > 50% response will be divided to two groups those with N2 disease or stage T4 will undergo two more cycles with induction TPF others will directly undergo treatment with RT (Total dose 70 Gy) in combination with cisplatin weekly (35mg/m2 ).Those who receive two more chemotherapy courses will be assessed clinically and by CT scan if no PD will continue to chemo and RT ,those with PD will undergo surgery Eight weeks following the completion of RT, patients will undergo a repeat direct laryngoscopy and a PET scan. The primary tumor site will be biopsied. Neck nodes that are persistent, clinically suspicious nodes, including PET positive nodes, will be biopsied. Patients with positive laryngeal biopsies following chemoradiation will undergo salvage surgery if possible supracricoid partial laryngectomy, otherwise laryngectomy. If the laryngeal biopsy is negative but clinically positive neck lymph nodes remain, patients will undergo neck nodal dissection.

Once patients are disease-free following chemoradiation and nodal neck dissections (if needed), patients will be followed every 6 weeks in the first year, followed by every 3 months in the second, every 6 month between 2 and 5 years. Patients whose physical examination or whose imaging studies are concerning for recurrent disease will undergo biopsy. If positive, they will undergo salvage laryngectomy.

Chemotherapy with Cisplatin, Docetaxel, and 5-Fluorouracil (TPF)

Docetaxel (Taxotere): Docetaxel 75 mg/m2 administered as an i.v. infusion over one hour on day #1.

With Docetaxel administration, all patients will receive dexamethasone 8 mg PO BID for 3 consecutive days, starting 1 day before docetaxel administration, or 10-20 mg IV on Day 1 prior to treatment with Docetaxel.

Cisplatin: Cisplatin 100 mg/m2, administered as an i.v. infusion will run over one hour on day #1 following docetaxel.

An aggressive antiemetic regimen is required before the administration of cisplatin, consisting of a serotonin antagonist, APREPITANT and a steroid.

5-Fluorouracil: 5-Fluorouracil 750 mg/m2 in 0.9% normal saline as a 24-hour continuous infusion, day's #1-4. The infusion will start after cisplatin administration.

Evaluation of Response to Treatment

Careful evaluation of tumor extent will be separately recorded for the primary tumor and regional nodes at specified intervals. These will be based on laryngoscopies performed pre-treatment, day 21 after start of induction chemotherapy, and 8 weeks after completion of chemoradiation. Standardized response criteria will be used. CT scans will be used at the discretion of the clinician to supplement clinical exams.

7.4.2 Biopsy of any persistent neck nodes is required if at the 8 week post -radiation evaluation is either clinical or radiologically positive. . Patients whose PET shows a CR at 8 weeks post will undergo clinical observation.

Diagnostic CT scans and/or PET scans will be obtained prior to scheduled endoscopies for tumor assessment. Post treatment a ct will be performed.

Outpatient clinical examinations will be performed at the completion of radiation therapy, at 6 week intervals during year 1 of follow-up,every 3 months during year 2 of follow-up, and 6-monthly during year 3 of follow-up. 8 Translational Studies

Tissue samples obtained at the time of laryngeal biopsies will be sent to laboratories for analysis of histologic growth pattern, p53 overexpression, Bcl-XL, Bcl-2 expression, HPV , EGFR expression, phosphorylated EGFR and stem cells levels . The tissue will be obtained during routine biopsies prior to the beginning of treatment, after completion of induction chemotherapy and after Radiation .the following techniques will be used: Immunohistochemistry, PCR and Western blot.

10 Response Assessment Criteria:

The patient's tumor will be tattooed by the surgeon,who will then measure the product of the longest primary tumor dimension and its perpendicular; following chemotherapy, the extent of the tumor will be measured for response. Treatment decisions (i.e. surgery vs Chemo+RT) are based on response of the tumor at the primary site.

Tumor responses to chemotherapy or chemoradiation will be determined clinically by the surgeon performing the DL.

Radiologic imaging studies will be used in conjunction with the physical examination in determining tumor response to chemotherapy or chemoradiation.

Clinical PR: Significant (>50%) reduction in the product of the longest primary tumor dimension and its perpendicular compared to pre-treatment clinical (endoscopic) measurements or imaging study as necessary.

Non-Responders (< PR): A 50% or less reduction in the product of the longest primary tumor dimension and its perpendicular compared to pre-treatment clinical (endoscopic) measurement or imaging study as necessary.

Criteria for Discontinuation of Treatment

1. Unacceptable adverse event(s).
2. Intercurrent illness, which prevents further administration of treatment.
3. Patient preference.
4. Progressive disease.
5. Life threatening or other unacceptable drug-related toxicity.
6. General or specific changes in the patient's condition that render the patient unacceptable for further treatment in the judgment of the investigators.

Radiation Therapy

13.1. General Considerations: All the patients in this study will receive either definitive radiotherapy or post operative irradiation. For those patients found to have a PR to induction therapy on repeat DL, definitive radiotherapy with Cisplatin will begin. Post operative radiation should begin as soon as adequate healing has been established. Usually, this will be within three to four weeks of the surgical procedure but must begin by six weeks.

13.2 Radiation Fields: The treatment volumes will be individual as for each patient depending upon the extent of disease. Tumor volumes will be outlined on the planning CT scans with the aid of pre-chemotherapy CT and, if available, PET scans, to ensure adequate irradiation of the pre-chemotherapy tumor volume. Treatment techniques will aim at adequate irradiation of the clinical and the sub-clinical disease. The therapy goals, specifying the intended doses to the primary tumor and lymph node metastases, and the intended doses to each lymph node level treated adjuvantly, will be detailed in the therapy chart. A CT-based display of the isodoses will be recorded, such that it will be feasible to assess whether the intended (prescribed) isodoses cover the targets adequately.

Doses:

Radiation with chemotherapy: Tumor doses will be expressed in Gy. The prescribed doses should encompass the targets. Treatment plans will be generated demonstrating adequate coverage of the target volume. The dose across the target volume should not vary by more than +/- 10% of the prescribed dose.The treatment will be given either using IMRT planning or 3D. Treatment will be given once daily, five days per week, two Gy per fraction to gross disease, and 1.6-2.0 Gy per fraction to subclinical disease. Total gross dose will be 70 Gy and subclinical disease dose will be 50-60 Gy.

Post Operative Radiation Therapy: The patient will be treated with conventional fractionation, 1.8-2.0 Gy per fraction, and five fractions per week in a continuous course. The dose to the tumor bed and lymph nodes will be 56-64 Gy, depending of the existence of extranodal extension or the existence of close surgical margins. Patients with gross residual disease or positive resection margins will receive total 66-70 Gy to the sites of residual disease.

Salvage Surgery

The extent of salvage surgery for either the primary tumor or regional nodes is dictated by the extent of the disease .

Salvage surgery may be required at the times of scheduled tumor assessments or any time tumor progression or recurrence is demonstrated by adequate biopsies of areas clinically suspicious for tumor involvement.

Primary site: Extent of surgery will vary between total laryngectomy and supracricoid subtotal laryngectomy in accordance with the inclusion and exclusion criteria specified).

Neck: Bilateral selective neck dissections will be performed in conjunction with salvage total laryngectomy for any patient initially staged N0 in the neck. Ipsilateral modified radical or radical neck dissection is required for any patient initially staged N+ who recurs or persists with cancer in that neck. At 8 weeks post radiation, neck dissection alone without laryngectomy is required for any patient with initial staging neck node > 3 cm in size who is PET positive or with biopsy proven palpable neck disease. 14.5

Informed Consent

All patients with stage III and IV squamous cell carcinoma of the larynx who are candidates for surgical resection will be screened for participation in this study.

.

Reporting Potentially Serious Adverse Events

Definitions

An adverse event is any new, undesirable medical experience or Change of an existing condition which occurs during or after treatment, whether or not considered product-related.

A serious adverse event is any untoward medical occurrence that

Suggests significant hazard or side effect that:

1. Results in death.
2. Is life-threatening (places the patient at immediate risk of death).
3. requires or prolongs inpatient hospitalization Is disabling or incapacitating.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed previously untreated, resectable, squamous cell carcinoma of the larynx.
* Disease must be Stage III or IV.
* Tumor must be potentially surgically resectable and curable with conventional surgery and radiation therapy.
* Patients must undergo pre-treatment endoscopic tumor staging and CT scanning of chest and neck.(pet scan optional)
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2.
* Pre-treatment laboratory criteria:

  * WBC > 3500/ul, granulocyte > 1500/ul.
  * Platelet count > 100,000/ul.
  * Calculated or measured creatinine clearance > 60 cc/min.
  * AST and ALT < 2.5 X ULN
* Patients must give documented informed consent to participate in this study.

Exclusion Criteria:

* Prior head and neck malignancy or active non-head and neck malignancy. Except for cured non-melanoma skin cancer,
* Prior head and neck radiation.
* Documented evidence of distant metastases.
* Active infection.
* Pregnancy or lactation. Patients must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Any medical or psychiatric illness which in the opinion of the principal investigator would compromise the patient's ability to tolerate this treatment.
* Age < 18 years.
* Patients with psychiatric/social situations that would limit compliance with study requirements are not eligible.
* Patients with Grade > 2 peripheral neuropathy.
* Any history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.

Criteria for supracricoid resection for chemo selection non responders

Inclusion Criteria :

* At least one functional arytenoids (physical and radiological examinations)
* Involvement of thyroid cartilage including extrathyroid cartilage extension.

Exclusion criteria:

* Subglottic extension anteriorly.
* Pre epiglottic extension.
* Subglottic extension laterally.
* Interarytenoid involvement.
* Two Arytenoids involved.

Criteria for supracricoid resection for Chemoradiation failure:

Inclusion Criteria:

* At least one functional arytenoid (physical and radiological examinations)
* Involvement of thyroid cartilage (with no radiological evidence for extra thyroid Extension).

Exclusion Criteria:

* Extrathyroid cartilage extension.
* Involvement preepiglottic space.
* Subglottic extension.
* Interarytenoid involvement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in larynx preservation free survival | 5 years

SECONDARY OUTCOMES:
Improvement in overall survival in patients treated under this regimen in comparison to historical control | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, MD, Principal Investigator — Rabin MC
Locations (1):
- Rabin MC, Petah Tikva, Israel